CLINICAL TRIAL: NCT01880801
Title: IMMUNOGLOBULINS ANTI PLATELETS IN BREAST MILK OF MATERNAL ITP
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Laniado Hospital (Other)
Responsible Party: Principal Investigator, Laniado Hospital, pediatric hemato-oncology, Laniado Hospital
Other Study IDs: 006-12-LND
Record Dates: First submitted 2013-06-17; First posted 2013-06-19 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2012-02

CONDITIONS: Mothers With ITP Condition
Keywords: ITP

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to determine whether mothers with Idiopathic thrombocytopenic purpura (ITP) has antibodies against platelets in breastfeeding milk aside control group of healthy mothers.

In order to prevent severe thrombocytopenia in infants born to mothers with ITP.

DETAILED DESCRIPTION:
Samples of breastfeeding milk and sera will be collected from 10 lactating women diagnosed with ITP and from 10 healthy women in the same stage after giving birth. Antibodies against platelets in the samples will be examined by using anti human IgM/G/A antibody following incubation of the serum/milk samples with platelets. The platelets will be from leftovers of samples send to platelets functionality test and found to be normal (the platelets samples will be taken without any identification and be marked only with lab number). The measurement will be done by flow cytometer. Sample will be consider as positive when the signal will be greater than 2 fold of control samples standard deviation. In addition, the presence of antibodies in different times from the birth will be checked in breastfeeding milk and sera of ITP patients. If the milk proteins and lipids will disturb the exam, the immunoglobulins from the milk will be isolated using Ig isolation kit from plasma.

ELIGIBILITY:
Inclusion Criteria:

* Maternal ITP
* Newborns above 35W and above 2.5 kg

Exclusion Criteria:

* mothers who do not breast feeding
* Thrombocytopenia from other reasons

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Lactating women diagnosed with ITP
Sampling Method: Probability Sample
Enrollment: 22 (Estimated)
Dates: Start 2013-08; Primary Completion 2014-08 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
IMMUNOGLOBULINS ANTI PLAITLETS IN BREST MILK OF MATERNAL ITP | 4 times in the first month after delivery

CONTACTS AND LOCATIONS:
Locations (1):
- Sharon Nechama, Laniado Hospital, Netanya, Israel, Israel